CLINICAL TRIAL: NCT01917227
Title: Evaluation of Group Health Teaching With Video in Diabetic Patients
Acronym: EGVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHIA-HUNG LIN, Department of Endocrinology and Metabolism, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 102-1452B
Record Dates: First submitted 2013-07-26; First posted 2013-08-06 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video (Experimental)
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video

SUMMARY:
Objective:Health videos and group education to allow patients to a correct understanding of diabetes and insulin treatment.

Method:

Standards and number of patients: The patients received subcutaneous insulin injection, estimated 30 people enrolled.

Experimental Design and Methods:

1. Screening out-patient treatment with insulin use, HbA1c> 8% or poor postprandial glucose (PPG)
2. At the time of the visits, invite the patient to participate in the Video group education on insulin therapy By answering some questions about insulin injections, such as: do not know how to perform; afraid of the pain; fear of inconvenience, give patients time to complete the questionnaire.

DETAILED DESCRIPTION:
Diabetes is a long-term chronic disease. The patients need to correct "knowledge and action" lifestyle in order to achieve effective blood glucose control. Upon the general control of diabetic patients in Taiwan, however, glycosylated hemoglobin (HbA1c) is not satisfactory. One of the important reasons is the low rate of insulin injection. For the use of insulin, the patient has many misconception. The patients in the clinic need to spend a lot of time to explain and description, but the results are not necessarily good. So we hope that in this part of the health education activities through organized groups Videos to assist doctors and patients as a bridge of communication, to enhance diabetes doctor thus contributing to glycemic control results.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent
2. Age over 20 years old
3. HbA1c>8% or PPG) > 200 mg/dl even under insulin therapy

Exclusion Criteria:

1. Vegetation status
2. Inability of visual or hearing contact with the video program

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-HUNG LIN, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan